CLINICAL TRIAL: NCT06544330
Title: A Phase 1, Open-Label Study to Evaluate the Safety and Tolerability of a Combination Autologous CD19 CAR T Cell Therapy (SYNCAR-001 + STK-009) in Subjects With Severe, Refractory Systemic Autoimmune Rheumatic Disease
Brief Title: A Phase 1 Study of SYNCAR-001 + STK-009 Without Conditioning Chemotherapy (Lymphodepletion) in Subjects With Severe, Refractory Systemic Autoimmune Rheumatic Disease
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Synthekine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STK-009-201
Record Dates: First submitted 2024-07-25; First posted 2024-08-09 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Systemic Lupus Erythematosus; Lupus Nephritis; Systemic Sclerosis
Keywords: CAR T; CD19-CAR T; Chimeric antigen receptor; IL-2
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SYNCAR-001 + STK-009 (Experimental): Dose escalation: A single fixed dose of autologous SYNCAR-001 CAR-T intravenously (IV) will be administered in combination with ascending doses of STK-009 subcutaneously (SC) in non-lymphodepleted patients.
  Dose expansion: A single fixed dose of autologous SYNCAR-001 CAR-T IV will be administered in combination with STK-009 SC at the RP2D in non-lymphodepleted patients.
  Interventions: Drug: SYNCAR-001; Drug: STK-009

INTERVENTIONS:
Drug: SYNCAR-001 — SYNCAR-001 is an autologous CD19-targeted CAR-T with co-expression of hoRb
Drug: STK-009 — STK-009 is a human orthogonal IL-2 cytokine selective for SYNCAR-001 CAR-T cells expressing hoRb

SUMMARY:
This is a phase 1 study of SYNCAR-001 + STK-009 in patients with severe, refractory systemic autoimmune rheumatic disease.

DETAILED DESCRIPTION:
SYNCAR-001 + STK-009 is a 2-component human orthogonal (ho) IL-2 receptor-ligand cell therapy consisting of (1) SYNCAR-001, a CD19-directed chimeric antigen receptor T cell (CAR-T) co-expressing an engineered IL-2 beta receptor (hoRb); and (2) STK-009, an engineered pegylated IL-2 cytokine (hoIL-2) selective for hoRb. This study is being conducted to evaluate the safety and efficacy of a single dose of SYNCAR-001 followed by multiple subcutaneously administered doses of STK-009. No conditioning chemotherapy (lymphodepletion) will be administered. The study will follow a 3+3 design during dose escalation followed by dose expansion at the recommended phase 2 dose (RP2D).

ELIGIBILITY:
General Inclusion Criteria:

Age ≥18 years at screening.

SLE Inclusion Criteria:

1. Clinical diagnosis of SLE according to the 2019 European League Rheumatism EULAR/ACR classification criteria.
2. Subject must be positive for at least one of the following at screening: Anti-dsDNA (above the upper limit of normal [ULN]); or anti-Sm (above the ULN); or anti-Chromatin (above the ULN).
3. Subjects with active, severe, non-renal SLE or subjects with active proliferative LN

SSc Inclusion Criteria:

1. Classified as SSc according to the ACR/EULAR classification criteria.
2. Diffuse cutaneous SSc (dcSSc) or SSc-associated ILD (SSc-ILD; significant or progressive).

General Exclusion Criteria:

1. History of or active central nervous system manifestations of autoimmune disease.
2. Prior treatment with anti-CD19 adoptive T cell therapy, or any prior gene therapy product (e.g., CAR T cell therapy).

SLE Exclusion Criteria:

1. Rapidly progressive glomerulonephritis.
2. End stage renal failure requiring dialysis or most recent renal biopsy with purely chronic lesions (Class III[C], IV-S[C], or IV-G[C]) if isolated renal disease.

SSc Exclusion Criteria:

1. FVC <50% of predicted or DLCO <40% of predicted.
2. Pulmonary arterial hypertension (PAH) requiring PAH-specific treatment.

Other protocol-defined criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2041-04 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities (DLTs) | Up to 28 days after SYNCAR-001 infusion
  Incidence of adverse events (AEs) meeting protocol defined DLT criteria in the dose escalation phase of the study.
Adverse Events | Up to 96 weeks after SYNCAR-001 infusion
  Incidence and severity of AEs including treatment-emergent AEs and serious AEs.

SECONDARY OUTCOMES:
Remission rate per Definition of Remission in SLE (DORIS) | Up to 96 weeks after SYNCAR-001 infusion
  For SLE only
Lupus Low Disease Activity State (LLDAS) attainment rate | Up to 96 weeks after SYNCAR-001infusion
  For SLE only
Change over time in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) | Up to 96 weeks after SYNCAR-001 infusion
  For SLE only. The SLEDAI-2K assessment consists of 24 items with a total score of 0 (no symptoms) to 105 (presence of all defined symptoms) with higher scores indicating increased disease activity.
Change over time in British Isles Lupus Activity Group (BILAG) score | Up to 96 weeks after SYNCAR-001 infusion
  For SLE only. The BILAG instrument assesses 97 clinical signs, symptoms, and laboratory parameters across 9 organ system domains related to SLE. BILAG scoring represents: A=severe disease, B=moderate disease, C=stable mild disease, D=inactive but previously active disease, E=never involved.
Change over time in levels of SLE and SSc serum autoantibodies | Up to 96 weeks after SYNCAR-001 infusion
Complete renal response rate (CRR) | Up to 96 weeks after SYNCAR-001 infusion
  Lupus Nephritis only. CRR will be defined as a UPCR < 0.5 and no eGFR decrease > 15% from baseline.
Change over time in Modified Rodnan Skin Score (mRSS) | Up to 96 weeks after SYNCAR-001 infusion
  Systemic Sclerosis only. mRSS measures skin thickness and is the sum of scores from 17 surface anatomic areas rated on a 0-3 scale (0=normal skin; 1=mild thickness; 2=moderate thickness; 3=severe thickness with inability to pinch the skin into a fold). mRSS ranges from 0 (best possible outcome) to 51 (worst possible outcome)
Proportion of subjects achieving revised Composite Response Index in Systemic Sclerosis (rCRISS-25) criteria | Up to 96 weeks after SYNCAR-001 infusion
  Systemic Sclerosis only. rCRISS-25 is the proportion of patients who improve in ≥ 2/5 ACR CRISS core items by 25% (except 5% for FVC) with no worsening of 1 core item
Proportion of subjects achieving rCRISS-25 criteria with no immunosuppressive therapy. | Up to 96 weeks after SYNCAR-001 infusion
  Systemic Sclerosis only
Change over time in pulmonary function tests | Up to 96 weeks after SYNCAR-001 infusion
  Systemic Sclerosis only. Pulmonary function tests include % predicted FVC (Forced Vital Capacity) and % predicted DLCO (Diffusing capacity of the lung for carbon monoxide)
Change over time in high resolution computed tomography of the chest for subjects with interstitial lung disease. | Up to 96 weeks after SYNCAR-001 infusion
  Systemic Sclerosis only. High resolution computed tomography images of the chest will be scored according to changes in interstitial lung disease using validated qualitative and quantitative methods

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Feinstein Institutes for Medical Research, Manhasset, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No